CLINICAL TRIAL: NCT00686322
Title: Phase IV Study of Concurrent Chemoradiotherapy With Paclitaxel and Cisplatin in Previously Untreated, Inoperable (Stage IIIa or IIIb) Non-small-cell Lung Cancer
Brief Title: Concurrent Chemoradiotherapy (CCRT) With Paclitaxel Plus Cisplatin in LA Non-small-cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-02-12
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2010-06

CONDITIONS: Non-small-cell Lung Cancer
Keywords: chemotherapy; radiotherapy; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Chemoradiotherapy; Paclitaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Induction one cycle of paclitaxel plus cisplatin (PC), concurrent 2 cycles of PC with radiotherapy, followed by 2 cycles of PC consolidation chemotherapy.
  Interventions: Drug: Concurrent chemoradiotherapy (paclitaxel plus cisplatin plus radiotherapy)

INTERVENTIONS:
Drug: Concurrent chemoradiotherapy (paclitaxel plus cisplatin plus radiotherapy) — Induction one cycle of paclitaxel plus cisplatin (PC), concurrent 2 cycles of PC with radiotherapy, followed by 2 cycles of PC consolidation chemotherapy.
  Other Names: paclitaxel; cisplatin

SUMMARY:
Present study is to investigate efficacy and toxicity profiles of induction one cycle of paclitaxel plus cisplatin (PC), concurrent 2 cycles of PC with radiotherapy, followed by 2 cycles of PC consolidation chemotherapy.

DETAILED DESCRIPTION:
Lung cancer is a major cause of cancer death in Taiwan and throughout the world in both developed and developing countries. More than 75% of NSCLC patients are inoperable because of either distantly metastatic disease or disease confined to one hemithorax with one or more criteria of unresectability at the time of presentation. The prognosis of such inoperable metastatic patients is poor.

The benefit of adding chemotherapy to radiation therapy for stage III disease of NSCLC is well-established. The largest of the prospective trials was sponsored by the Radiation Therapy Oncology Group (RTOG), ECOG, and the Southwest Oncology Group (SWOG), and allocated 490 patients to receive 2 months of cisplatin + vinblastine chemotherapy followed by 60 Gy of radiation at 2 Gy per fraction; or one of two radiation-alone arms. Overall survival was statistically superior for the patients receiving chemotherapy and radiation versus the other two arms of the study (13.2 months vs 12 months, vs 11.4 months, respectively; p=0.04).

Administration of chemotherapy concurrently with radiation therapy theoretically improves local control by sensitizing the tumor to radiation, while simultaneously treating systemic disease, albeit at the expense of greater local toxicity. Two large phase III studies suggest improvement in both local control and survival with concurrent chemoradiotherapy as compared with sequential chemotherapy followed by radiation for patients with stage III NSCLC. Although rates of nonhematologic toxicity were higher on the concurrent arms, median survival time trended toward superiority in the concomitant chemotherapy plus daily radiation arm compared with the sequential arm.

One source of debate is whether the addition of induction or consolidation chemotherapy adds anything to concomitant chemoradiotherapy, with numerous intergroup trials underway. CALGB has completed a randomized phase II study of two cycles of induction chemotherapy followed by two additional cycles of the same drugs with concomitant radiotherapy. The three treatment arms included four cycles of cisplatin (80 mg/m2) combined with either gemcitabine, paclitaxel, or vinorelbine. Radiotherapy was completed during the last two cycles to a total of 66 Gy. Response rates were similar, and median survival for all patients was 17 months with no clearly superior arm evident in this randomized phase II trial.

We proposed this clinical trial to evaluate the efficacy and toxicity profile of combination chemotherapy with paclitaxel and cisplatin in previously untreated, stage IIIa/IIIb NSCLC patients who received 1 cycle of induction chemotherapy, followed by concurrent chemoradiotherapy, with 2 cycles of consolidation chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytological diagnosis of inoperable locally advanced (stage III) NSCLC.
* No prior chemotherapy, immunotherapy, or radiotherapy.
* Performance status of 0 to 2 on the Zubrod scale.
* Clinically measurable disease, defined as bidimensionally measurable lesions with clearly defined margins on x-ray, scan, or physical examination. Lesions serving as measurable disease must be at least 1 cm by 1 cm, as defined by computerized tomography (CT) scan, magnetic resonance imaging (MRI), or chest x-ray.
* Estimated life expectancy of at least 12 weeks.
* Patient compliance and geographic proximity that allow adequate follow-up.
* Adequate bone marrow reserve: white blood cell (WBC) count *4,000/mm3, platelets >100,000/mm3, and hemoglobin *10 g/dL.
* Informed consent from patient.
* Males or females 18 years of age or older.
* If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine contraceptive device [IUD], birth control pills, or barrier device) during and for three months after trial.

Exclusion Criteria:

* Active infection (at the discretion of the investigator).
* Inadequate liver function (total bilirubin >1.5 times above normal range); alanine transaminase (ALT) and aspartate transaminase (AST) greater than 3 times normal (ALT and AST may be elevated to 5 times normal in patients with known metastatic disease in the liver).
* Inadequate renal function (creatinine >2.0 mg/dL).
* Pregnancy or not using appropriate birth control during the study.
* Breast feeding.
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Use of any investigational agent in the month before enrollment into the study.
* Patients with leukemia and/or a secondary primary carcinoma except for patients who have had curative therapy to basal cell carcinoma.
* Concomitant myelosuppressive radiotherapy, chemotherapy, hormonal therapy, or immunotherapy will not be allowed except as previously noted for radiation.
* Active cardiac disease requiring therapy for failure, angina, and/or arrhythmias; infarctions within the preceding six months (exception: any patient whose cardiac failure is compensated on medications).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of this treatment modality in patients with inoperable stage III NSCLC | one year

SECONDARY OUTCOMES:
To determine the toxicity profiles of this treatment modality in patients with inoperable stage III NSCLC | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Min Chen, MD, PhD., Principal Investigator — Chest Department, Taipei VGH
Locations (1):
- Taipei VGH, Taipei, Taiwan